CLINICAL TRIAL: NCT05008744
Title: Laser Photocoagulation of Communicating Vessels in Twin-to-Twin Transfusion Syndrome (TTTS)
Brief Title: Laser Photocoagulation of Communicating Vessels in Twin-to-Twin Transfusion Syndrome
Status: Recruiting | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Martin Walker, Co-Director Seattle Childrens Fetal Intervention and Surgery Program, Clinical Assistant Professor, Seattle Children's Hospital
Other Study IDs: 00003168
Record Dates: First submitted 2021-07-21; First posted 2021-08-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Twin to Twin Transfusion as Antepartum Condition; Monochorionic Diamniotic Placenta
Keywords: Twin; Monochorionic; Fetoscopy; Laser

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Amniotic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients presenting with TTTS: Pregnant persons between 16 and 36 weeks of pregnancy with a diagnosis of twin to twin transfusion syndrome
  Interventions: Procedure: Fetoscopic laser ablation

INTERVENTIONS:
Procedure: Fetoscopic laser ablation — Under ultrasound guidance, a 2 mm skin incision will be made and a 10Fr Cook Check Flow valve cannula and trocar will be introduced into the amniotic cavity.
  The communicating vessels will be located endoscopically using a Storz straight or curved semirigid fetoscopes in a fetoscopic sheath, a Humanitarian Use Device, used with permission of the Federal Drug Administration under a Humanitarian Device Exemption agreement with Karl Storz, Inc, and will be ablated with a diode laser fiber that is passed through the operating channel of the endoscope.

SUMMARY:
The purpose of this study is to evaluate the use of diode laser photocoagulation of the communicating vessels in twin-to- twin transfusion syndrome (TTTS) with respect to maternal, fetal and neonatal outcomes.

DETAILED DESCRIPTION:
Patients will undergo an intake evaluation followed by a detailed ultrasound examination to rule out the presence of congenital anomalies and to assess the hemodynamic status of the fetuses and any pre-existing cerebral damage. The following data will be collected, as is identical to the standard of care in evaluating monochorionic twins

Maternal

* Age
* Gravidity and parity
* BMI
* Race/ethnicity
* Gestational age
* The presence of any symptoms
* Cervical length

Fetal

* Estimated fetal weight
* Detailed anatomy
* Doppler evaluation of umbilical cord, ductus venosus and middle cerebral arteries
* Evaluation of the myocardial performance indices
* Amniotic fluid volume
* Placental position
* Cord insertions

Patients will then be counseled about the risks and benefits of the procedure and will be asked to sign an informed consent.

The procedure will be performed under a spinal or local anesthesia at the discretion of the anesthesiologist and surgeon based upon placental position, maternal hemodynamic stability and maternal anxiety and ability to cooperate. Ultrasound guidance will help to select an appropriate incisional site. Under ultrasound guidance, a 2 mm skin incision will be made and a 10 French Cook Check Flow valve cannula and trocar will be introduced into the amniotic cavity. An amniotic fluid sample will be obtained and sent for microbiological studies. A small aliquot of fluid will also be set aside for future institutional review board approved studies (see detail regarding banking below).

The communicating vessels will be located endoscopically using a Storz straight or curved semirigid fetoscopes in a fetoscopic sheath, a Humanitarian Use Device, used with permission of the Federal Drug Administration under a Humanitarian Device Exemption agreement with Karl Storz, Inc, and will be ablated with a diode laser fiber that is passed through the operating channel of the endoscope. The Laser used is a Dornier Diode laser using a power of 30-40 Watts. At the conclusion of the anastomotic ablation, an ablation line will be created across the vascular equator, effectively dichorionizing the placenta. The procedure will be monitored both endoscopically and sonographically. The presence of fetal heart activity will be documented at the beginning and end of the procedure. An amniodrainage of the larger sac will be performed at the conclusion of the procedure to leave the amniotic fluid volume of that sac at a normal level.

ELIGIBILITY:
Inclusion Criteria:

* Single placenta (Monochorionic)
* Polyhydramnios present in recipient twin (Greater than 8 cm maximum vertical pocket below 20 weeks and greater than a 10 cm pocket for greater than 20 weeks gestational age)
* Oligohydramnios present in donor twin (Less than 2 cm maximum vertical pocket)
* Prominent bladder in the recipient/ non-filling bladder in the donor
* Thin dividing membrane

Exclusion Criteria:

* Patients unwilling to participate in the study or to be followed up
* Presence of major congenital anomalies incompatible with survival
* Active pre-term labor Ruptured membranes
* Chorioamnionitis
* Vaginal bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant persons presenting with a diagnosis of twin to twin transfusion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2031-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Survival | Immediately after the surgery to discharge from the hospital after delivery
  Survival to discharge from the nursery of affected babies

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Walker, MD, Principal Investigator — Seattle Childrens Hospital
Locations (2):
- United States (2):
  - Seattle Childrens Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
No sharing planned